CLINICAL TRIAL: NCT01671332
Title: Randomized Phase II Study of Suramin and Docetaxel Versus Docetaxel in Non-Small Cell Lung Cancer After Failure of First-Line Chemotherapy
Brief Title: Docetaxel +/- Suramin in 2nd Line Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Medical College of Wisconsin (Other); Optimum Therapeutics, LLC (Industry); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO11508; A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison); 2012-0118 (Other: Institutional Review Board); NCI-2012-01113 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2012-06-25; First posted 2012-08-23 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Carcinoma, Non Small Cell Lung
Keywords: Carcinoma, non small cell lung; Second line; Third line
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Suramin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel
- Docetaxel plus Suramin (Experimental)
  Interventions: Drug: Suramin; Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — IV over 60 minutes, 75 mg/m2
  Other Names: Taxotere
  Arms: Docetaxel
Drug: Suramin — IV over 30 minutes
  Arms: Docetaxel plus Suramin
Drug: Docetaxel — IV over 60 minutes. 56 mg/m2
  Other Names: Taxotere
  Arms: Docetaxel plus Suramin

SUMMARY:
The overall purpose of the study is to determine whether or not the inclusion of suramin to standard treatment with docetaxel improves progression-free survival for patients with advanced non-small cell lung cancer in the second and third line settings.

DETAILED DESCRIPTION:
The overall purpose of the study is to determine whether or not the inclusion of suramin to standard treatment with docetaxel improves progression-free survival for patients with advanced non-small cell lung cancer in the second and third line settings.

Secondary objectives include:

* To compare response rate of patients in both treatment arms
* To compare overall survival of patients in both treatment arms
* To compare toxicity in both treatment arms
* To determine whether the survival benefit from suramin is associated with reduced M-phase entry in peripheral blood lymphocytes

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of non-small cell lung cancer
* Documented disease progression after first-line chemotherapy for non-small cell lung cancer
* Stable and treated CNS metastasis is allowed
* Radiation must be completed at least 2 weeks prior to starting protocol treatment
* Major surgery must be completed at least 4 weeks prior to starting protocol treatment
* ECOG performance status 0-2
* Sexually active patients must use adequate contraception
* Adequate bone marrow function
* Adequate renal function
* Adequate liver function

Exclusion Criteria:

* Severe hypersensitivity reaction to docetaxel
* Pre-existing grade 3 or 4 neuropathy
* Women who are pregnant or breastfeeding
* Uncontrolled intercurrent illness
* Receipt of 3 or more prior chemotherapy regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2015-06-11 (Actual); Study Completion 2016-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Traynor, MD, Principal Investigator — University of Wisconsin, Madison; Rafael Santana-Davila, MD, Study Chair — Medical College of Wisconsin
Locations (2):
- United States (2):
  - University of Wisconsin Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from June 2012 through April 2014.
Groups:
- Docetaxel: Docetaxel: IV over 60 minutes, 75 mg/m2
  Participants with disease progression on the docetaxel arm were allowed to cross over to the suramin arm.
Period: Overall Study
Arm/Group | Docetaxel | Docetaxel Plus Suramin
Started | 40 | 40
Crossed Over to Docetaxel Plus Suramin (Participants with disease progression on Docetaxel Arm were allowed to crossover to Suramin.) | 0 | 13 (Participants with disease progression on Docetaxel Arm were allowed to crossover to Suramin.)
Completed | 39 | 39
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel | Docetaxel Plus Suramin | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Customized [Number; unit: participants]
  18-39 years | 0 | 0 | 0
  40-49 years | 1 | 2 | 3
  50-59 years | 18 | 11 | 29
  60-69 years | 17 | 16 | 33
  70-79 years | 3 | 9 | 12
  80-89 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 22 | 35
  Male | 27 | 18 | 45
Race/Ethnicity, Customized [Number; unit: participants]
  White, Not of Hispanic Origin | 38 | 35 | 73
  Black or African American, Not of Hispanic Origin | 2 | 2 | 4
  Hispanic or Latino | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival in Months
Description: Compare progression-free survival (PFS) in participants with advanced NSCLC treated with docetaxel with or without suramin after failure of first-line chemotherapy. PFS is defined as the duration of time from the time of randomization to time of disease progression or death, whichever occurs first.
Time Frame: Up to 1 year
Population: The 13 participants that crossed over to the Docetaxel plus Suramin arm did so after progressing on the standard arm. Their progression-free survival was therefore purely determined by the arm of randomization and not influenced by the cross-over.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel | Docetaxel Plus Suramin
Number analyzed (Participants) | 40 | 40
months | 2.8 [0.9 to 4.2] | 1.6 [1.4 to 2.1]

2. Secondary Outcome: Response Rate Per RECIST 1.1 Criteria
Description: Response rate per RECIST 1.1, as follows:
  Complete response (CR): Disappearance of all extranodal target lesions. All pathological lymph nodes must have decreased to <10 mm in short axis Partial response (PR): At least 30% decrease in the sum of longest diameters (SLD) of target lesions, taking as reference the baseline sum diameters Progressive disease (PD): SLD increased by at least 20% from the smallest value on study (including baseline, if that is smallest). The SLD must also demonstrate an absolute increase of at least 5 mm. (Two lesions increasing from 2mm to 3mm, for example, does not qualify).
  Stable disease (SD): Neither sufficient shrinkage to qualify for PR not sufficient increase to qualify for PD
Time Frame: Up to 1 year
Population: The 13 participants that crossed over to the Docetaxel plus Suramin arm did so after progressing on the standard arm. Their response rate was determined by the arm of randomization and not influenced by the cross-over.
Measure: Number; unit: participants
Arm/Group | Docetaxel | Docetaxel Plus Suramin
Number analyzed (Participants) | 40 | 40
participants
  Partial Response | 1 | 3
  Stable Disease | 17 | 11
  Progressive Disease | 17 | 25
  Not Assessed | 5 | 1

3. Secondary Outcome: Overall Survival
Description: Compare overall survival of participants in both treatment arms.
Time Frame: Up to 50 months
Population: The 13 participants that crossed over did so after progressing on the standard arm. The overall survival was determined for the arm of randomization without regard of cross-over. Cross-over was provided as option for participants to have the possible benefit of the new treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel | Docetaxel Plus Suramin
Number analyzed (Participants) | 40 | 40
months | 5.3 [5.0 to 8.0] | 4.1 [3.2 to 7.6]

4. Secondary Outcome: Number of Participants With Toxicity/Adverse Events From Treatment
Description: The investigators will compare the toxicity profiles of the two arms of therapy to determine if the docetaxel + suramin has a more favorable toxicity profile than docetaxel alone. This count includes only adverse events considered definitely, probably, or possibly due to treatment.
Time Frame: Up to 2 years
Population: The 13 participants that crossed over did so after progressing on the standard arm. Reported here are the number of participants who experienced adverse events on the arm of randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel | Docetaxel Plus Suramin
Number analyzed (Participants) | 40 | 40
Participants | 35 | 31

5. Secondary Outcome: Evaluation of Peripheral Blood Lymphocytes for DNA Damage-induced Checkpoint Control.
Description: The investigators hypothesize that suramin in combination with docetaxel improves response rates and survival by increasing the cancer cell population in the M phase of the cell cycle. The G2-M checkpoint control score, defined as (%M-phase arrested cells after cisplatin+suramin)/(%M-phase arrested cells after cisplatin), is an indicator of the effect of suramin on cell accumulation in the M-phase. G2-M checkpoint control was evaluated as a predictor of PFS and OS in participant receiving suramin by linear correlation.
Time Frame: Baseline
Population: All participants who yielded good quality PBL samples were included.
Measure: Mean (Standard Deviation); unit: G2-M checkpoint control score
Arm/Group | Docetaxel | Docetaxel Plus Suramin
Number analyzed (Participants) | 18 | 28
G2-M checkpoint control score | 0.91 (0.37) | 1.30 (0.89)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from on-study through 30 days after last treatment dose, or until resolution/ stabilization of AEs occurred if longer than 30 days.
Description: AEs are reported by toxicity category. All Cause Mortality includes death greater than 30 days after the subject's off treatment date. SAEs and AEs are reported for all participants randomized to the Docetaxel arm (N=40), and all participants both randomized (N=40) and crossed over to (N=13) to the Docetaxel and Suramin arm, for a total of N=53.
Arm/Group | Docetaxel | Docetaxel Plus Suramin
All-Cause Mortality (participants affected / at risk) | 40/40 | 37/40
Serious Adverse Events (participants affected / at risk) | 19/40 | 26/53
Other Adverse Events (participants affected / at risk) | 39/40 | 49/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (N=40) | Docetaxel Plus Suramin (N=53)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Death NOS (General disorders) | 3 (3) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Esophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Febrile neutropenia (Cardiac disorders) | 2 (3) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
INR increased (Investigations) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 2 (2)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Peripheal ischemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (2)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thromboembolic Event (Vascular disorders) | 3 (3) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle Weakness Right-Sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (N=40) | Docetaxel Plus Suramin (N=53)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 8 (9)
Anemia (Blood and lymphatic system disorders) | 8 (9) | 14 (15)
Anorexia (Metabolism and nutrition disorders) | 6 (8) | 10 (10)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 5 (5)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Blood any lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
CPK increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Death NOS (General disorders) | 2 (2) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 7 (8)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 3 (4)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 11 (13)
Edema limbs (General disorders) | 4 (4) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Fatigue (General disorders) | 18 (24) | 22 (35)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Fever (General disorders) | 3 (3) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 2 (3)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (7)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 7 (8)
Hypertension (Vascular disorders) | 4 (7) | 4 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (5) | 6 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 7 (9)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Infusion related reaction (General disorders) | 1 (1) | 1 (1)
INR increased (Investigations) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (3)
Lung infection (Infections and infestations) | 4 (4) | 1 (2)
Lymphocyte count decreased (Investigations) | 9 (26) | 9 (18)
Malaise (General disorders) | 0 (0) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1) | 6 (6)
Mucositis oral (Gastrointestinal disorders) | 6 (6) | 6 (6)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (9) | 10 (12)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 16 (27) | 8 (16)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 5 (9) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peripheral motor neurpathy (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (11) | 6 (8)
Pharyngitis (Infections and infestations) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (4) | 2 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (4)
Watering eyes (Eye disorders) | 2 (3) | 1 (4)
White blood cell decreased (Investigations) | 16 (27) | 10 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less